CLINICAL TRIAL: NCT02720588
Title: Investigating Neuroimaging Endophenotypes for Autism Spectrum Disorder
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201505142RINC
Record Dates: First submitted 2016-03-22; First posted 2016-03-28 (Estimated); Last update posted 2021-09-02 (Actual); Status verified 2021-09

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- ASD group: Subjects have a clinical diagnosis of autistic disorder or Asperger disorder defined by the DSM-IV criteria
- Sibling group: Sex-matched unaffected siblings of ASD probands
- TD group: Typically developing controls without lifetime ASD or a family history of ASD

SUMMARY:
Specific Aims: This study aims to examine the hypothesis that individuals with Autism spectrum disorder (ASD) and their unaffected siblings shared alterations in gray and white matter volume and their associated intrinsic functional connectivity, to build upon limited literature about neuroimaging endophenotypes of ASD. The investigators also aim to test whether these shared differences are associated with behavioral autistic traits.

DETAILED DESCRIPTION:
Autism spectrum disorder (ASD) is a highly heritable neurodevelopmental disorder, yet the search for genes with a definitive role in its etiology has remained elusive. Deconstructing the disorder with endophenotypic approach should boost the statistical power of genetic studies and clarify the pathophysiology of autism. Neuroimaging data provides evidence for atypical trajectories of brain growth in ASD, which result in differences in neuroanatomy and connectivity in the widespread neural systems. As genetic factors are responsible for a significant amount of variation in neuroanatomy and intrinsic functional connectivity, shared alterations in brain morphology and associated functional connectivity between individuals with ASD and their unaffected siblings is likely a useful endophenotype. Nonetheless, such multi-modal approach has never been tested in study on endophenotypic markers for ASD. The study aims to fill in the gap.

The investigators plan to recruit 90 participants (30 adults with ASD, 30 unaffected siblings, and 30 healthy controls), without current and past history of any systemic physical illness, neither any major psychiatric disorder other than ASD. All the participants will receive psychiatric interviews (the Chinese version of the Autism Diagnostic Interview-Revised, ADI-R; the Chinese Version of the Kiddie Epidemiologic version of the Schedule for Affective Disorders and Schizophrenia, K-SADS-E). They will receive the Wechsler Adult Intelligence Scale-3rd edition(WAIS-III) first to ensure their full-scale IQ greater than 70. The MRI assessments (T1 imaging, single-echo echo planar imaging(EPI) resting-state fMRI) will be subsequently arranged within 2 weeks after psychiatric/neuropsychological assessments.

The investigators anticipate that this study (1) will be the first report in Taiwan to report neuroimaging endophenotypes for ASD; (2) will be the first report in the world on the shared structural and functional connective differences by ASD and their unaffected siblings; (3) will provide further evidence about the mechanism underpinning the broad autism phenotype.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who have a clinical diagnosis of autistic disorder or Asperger disorder defined by the DSM-IV criteria

Exclusion Criteria:

1. Systemic medical illness
2. Current symptoms or lifetime history of DSM-5 diagnosis of mood disorder, any psychotic disorder, substance use disorder, learning disorder, anxiety disorder, claustrophobia, obsessive compulsive disorder, or mental retardation.
3. With neurodegenerative disorder, epilepsy, involuntary movement disorder, congenital metabolic disorder, brain tumor, history of severe head trauma, and history of craniotomy;
4. Full-scale IQ < 70.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: The sample consists of 30 adults with ASD, and 30 sex-matched unaffected siblings, and 30 healthy volunteers.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Psychiatric Interview | 1 hour
  Subjects will be interviewed by Chinese Version of the Kiddie Epidemiologic version of the Schedule for Affective Disorders and Schizophrenia (K-SADS-E)

CONTACTS AND LOCATIONS:
Overall Officials: Hsiang-Yuan Lin, MD, Principal Investigator — Dept of Psychiatry, National Taiwan University Hospital; Susan Shur-Fen Gau, MD, PhD, Study Director — National Taiwan University Hospital & College of Medicine
Locations (1):
- National Taiwan Univeristy Hospital, Taipei, Taiwan